CLINICAL TRIAL: NCT07234916
Title: The Impact of Multivitamin Supplementation on Micronutrient Levels in GLP-1 Users: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Multivitamin Impact on Micronutrient Status in GLP-1 Users: A Randomized Trial
Acronym: VITAGLP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: weightworks Clinic (Unknown)
Responsible Party: Principal Investigator, Bart Torensma, Clinical epidemiologist, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLP-1-RCT-2025; ABR 2025 GLP (Other: The Netherlands Medical Research Portal (CCMO))
Record Dates: First submitted 2025-04-25; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Weight Loss; Nutritional Deficiencies; GLP - 1; Obese Patients
Keywords: weightloss; obesity; GLP-1; Nutritional deficiencies
MeSH Terms: conditions — Weight Loss; Malnutrition; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Multivitamin Supplementation) (Experimental): Participants in this group will receive a daily multivitamin supplement formulated to provide comprehensive micronutrient support. The supplement will be taken once daily with a meal for the 12-month intervention period following randomization.
  Interventions: Dietary Supplement: Multivitamin Supplementation
- Group B (Placebo) (Placebo Comparator): Participants in this group will receive a matching placebo that is identical in appearance, taste, and packaging to the active multivitamin supplement. The placebo will be taken once daily with a meal for the 12-month intervention period following randomization.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Multivitamin Supplementation — Multivitamin Supplementation
  Arms: Group A (Multivitamin Supplementation)
Other: Placebo — Placebo vitamine
  Arms: Group B (Placebo)

SUMMARY:
Rationale: Glucagon-Like Peptide-1 (GLP-1) receptor agonists have emerged as effective treatments for obesity and associated medical conditions. However, patients may be at risk of micronutrient deficiencies during therapy due to reduced appetite, altered gastrointestinal physiology, and weight loss. Multivitamin supplementation is commonly prescribed to mitigate these risks, but the necessity and efficacy of multivitamin use in GLP-1 users remain debatable, as some clinicians advocate for routine supplementation while others do not.

Objective: To assess the differences in micronutrient levels between patients who use multivitamin supplements while on GLP-1 therapy and those who do not, to provide evidence on the necessity and benefits of supplementation.

Study Design: Randomized, double-blind, placebo-controlled trial. Study Population: Adults with obesity (BMI ≥30 kg/m² or ≥27 kg/m² with obesity-associated medical problems) currently using GLP-1 receptor agonists for at least 3 months with stable dosing.

Intervention:

* Group A (Intervention): Multivitamin supplementation while on GLP-1 therapy
* Group B (Control): Matching placebo while on GLP-1 therapy Main Study Parameters/Endpoints: The primary outcomes are the differences in serum levels of Vitamin B12, Vitamin D, and Ferritin between the multivitamin and placebo groups after 12 months of supplementation while on GLP-1 therapy.

Nature and Extent of the Burden and Risks: Participants will undergo blood sampling at four timepoints: baseline (before starting GLP-1 therapy), at randomization (3 months of stable GLP-1 therapy), and at 6 and 12 months post-randomization. The risks associated with the study are minimal and primarily related to blood sampling and potential side effects of multivitamin supplementation. The burden includes time commitment for study visits and daily supplement intake.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 to 70 years.
* Start with the use of Tirzepatide GLP-1 receptor agonists and for at least 3 months with stable dosing before randomization.
* BMI ≥30 kg/m² or ≥27 kg/m² with obesity-associated medical problems (such as type 2 diabetes, hypertension, or dyslipidemia) at the start of GLP-1 therapy
* Willing and able to provide informed consent
* Able to comply with study procedures and follow-up visits
* Own vitamins should be completely discontinued 2 weeks before the start

Exclusion Criteria:

* Known allergy or hypersensitivity to any components of the multivitamin supplement
* Current use of other vitamin or mineral supplements
* Pregnancy or planning pregnancy during the study period
* Patients who follow a vegan diet.
* Active malignancy or ongoing cancer treatment
* Severe kidney disease (eGFR <30 mL/min/1.73m²)
* Severe liver disease (Child-Pugh C)
* History of metabolic bariatric surgery
* Participation in other clinical trials within the past 3 months
* Any condition that, in the investigator's opinion, would interfere with study participation or compromise patient safety

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2027-03-16 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
serum levels | 15 months
  1. Vitamin B12 (Reference range: 200-500 pmol/L)
  2. Vitamin D (Reference range: 50-200 nmol/L)
  3. Ferritin (Reference range: 30-388 μg/L)
  4. Folic acid (Reference range: 10-45 nmol/L)

SECONDARY OUTCOMES:
other micronutrient levels | 12 months
  Changes in other micronutrient levels from baseline to 12 months, including:
  * Iron (10-30 μmol/L)
  * Vitamin B1 (70-180 nmol/L)
  * Vitamin B6 (35-110 nmol/L)
  * Zinc (10-18 μmol/L)
  * Magnesium (0.70-1.05 mmol/L)
  * Calcium:
  Total serum calcium: 2.15-2.55 mmol/L) Ionized calcium: 1.16-1.32 mmol/L PTH (Parathyroid Hormone) (1.6-6.9 pmol/L)
  Changes in additional iron-related functional markers:
  * Transferrin (2.0-3.6 g/L)
  * Transferrin saturation (20-45%)
  * Total iron binding capacity 2. Changes in hematological parameters:
  * Hemoglobin (Female: 7.5-10.0 mmol/L; Male: 8.5-11.0 mmol/L)
  * Mean Corpuscular Volume (MCV) (80-100 fL)
  * HbA1c (4.0-6.0% (20-42 mmol/mol)) Inflammation and protein status
  * C-reactive protein (CRP): <10 mg/L
  * Albumin: 35-50 g/L Incidence of clinically significant deficiencies requiring intervention Correlation between weight loss parameters (%TWL, %EWL) and changes in micronutrient levels

OTHER OUTCOMES:
Weight loss | 12 months
  Weight and BMI changes throughout the study period
GLP adherence | 12 months
  Adherence to GLP-1 therapy and study medication
diet | 12 months
  Dietary intake patterns (assessed through food frequency questionnaires)
QoL | 12 months
  Quality of life measures
Body composition assessment | 12 months
  * Measured at baseline, 6 months, and 12 months
  * Parameters: fat mass, fat-free mass, muscle mass, visceral fat
Resting Energy Expenditure (REE) | 12 months
  Measured via indirect calorimetry

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - WeightWorks Clinics, Amersfoort
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
The investigator will be responsible for the data analysis. The analysis will be performed on a blinded data set after medical/scientific review has been completed, all protocol violations have been identified, and the data set has been declared complete. All data will be collected in a data management system (Castor EDC, Amsterdam, The Netherlands; https://www.castoredc.com) and performed according to Good Clinical Practice guidelines, Data Protection Directive certificate and complies with Title 21 CFR Part 11. Furthermore, the datacenter where all the research data is stored is ISO27001, ISO9001 certified and the Dutch NEN7510 certified.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Bettadapura S, Dowling K, Jablon K, Al-Humadi AW, le Roux CW. Changes in food preferences and ingestive behaviors after glucagon-like peptide-1 analog treatment: techniques and opportunities. Int J Obes (Lond). 2025 Mar;49(3):418-426. doi: 10.1038/s41366-024-01500-y. Epub 2024 Mar 7. PMID 38454010
- [Result] Friedrichsen M, Breitschaft A, Tadayon S, Wizert A, Skovgaard D. The effect of semaglutide 2.4 mg once weekly on energy intake, appetite, control of eating, and gastric emptying in adults with obesity. Diabetes Obes Metab. 2021 Mar;23(3):754-762. doi: 10.1111/dom.14280. Epub 2021 Jan 3. PMID 33269530
- [Result] Mechanick JI, Butsch WS, Christensen SM, Hamdy O, Li Z, Prado CM, Heymsfield SB. Strategies for minimizing muscle loss during use of incretin-mimetic drugs for treatment of obesity. Obes Rev. 2025 Jan;26(1):e13841. doi: 10.1111/obr.13841. Epub 2024 Sep 19. PMID 39295512
- [Result] He L, Li Q, Yang Y, Li J, Luo W, Huang Y, Zhong X. Pharmacovigilance study of GLP-1 receptor agonists for metabolic and nutritional adverse events. Front Pharmacol. 2024 Jul 8;15:1416985. doi: 10.3389/fphar.2024.1416985. eCollection 2024. PMID 39040467
- [Result] Liu L, Chen J, Wang L, Chen C, Chen L. Association between different GLP-1 receptor agonists and gastrointestinal adverse reactions: A real-world disproportionality study based on FDA adverse event reporting system database. Front Endocrinol (Lausanne). 2022 Dec 7;13:1043789. doi: 10.3389/fendo.2022.1043789. eCollection 2022. PMID 36568085
- [Result] Sargeant JA, Henson J, King JA, Yates T, Khunti K, Davies MJ. A Review of the Effects of Glucagon-Like Peptide-1 Receptor Agonists and Sodium-Glucose Cotransporter 2 Inhibitors on Lean Body Mass in Humans. Endocrinol Metab (Seoul). 2019 Sep;34(3):247-262. doi: 10.3803/EnM.2019.34.3.247. PMID 31565876
- [Result] Gentinetta S, Sottotetti F, Manuelli M, Cena H. Dietary Recommendations for the Management of Gastrointestinal Symptoms in Patients Treated with GLP-1 Receptor Agonist. Diabetes Metab Syndr Obes. 2024 Dec 19;17:4817-4824. doi: 10.2147/DMSO.S494919. eCollection 2024. PMID 39722834
- [Result] Christensen S, Robinson K, Thomas S, Williams DR. Dietary intake by patients taking GLP-1 and dual GIP/GLP-1 receptor agonists: A narrative review and discussion of research needs. Obes Pillars. 2024 Jul 25;11:100121. doi: 10.1016/j.obpill.2024.100121. eCollection 2024 Sep. PMID 39175746
- [Result] Moiz A, Filion KB, Tsoukas MA, Yu OH, Peters TM, Eisenberg MJ. Mechanisms of GLP-1 Receptor Agonist-Induced Weight Loss: A Review of Central and Peripheral Pathways in Appetite and Energy Regulation. Am J Med. 2025 Jun;138(6):934-940. doi: 10.1016/j.amjmed.2025.01.021. Epub 2025 Jan 31. PMID 39892489